CLINICAL TRIAL: NCT02037763
Title: A Prospective Controlled Trial to Identify Biomarkers Involved in the Transition From Acute to Persistent Chronic Low Back Pain
Brief Title: A Prospective Trial to Identify Biomarkers Involved in the Transition From Acute to Persistent Chronic Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Parma (Other)
Collaborators: GENOS (Other); Ip Research Consulting Sasu (Industry); Helmholtz Zentrum München (Industry); YURII AULCHENKO (Unknown); King's College London (Other)
Responsible Party: Principal Investigator, Massimo Allegri, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: Pain-OMICS PRT
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Acute Low Back Pain; Chronic Low Back Pain
Keywords: Low back pain; GWAS; Glycomics; Activomics; Epigenetics
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be collected at recruitment in all enrolled patients. Blood samples will be collected also at the 3 months and 6 months follow up visits in patients who will develop CLBP after the episode of acute LBP.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective observational cohort multinational clinical study. There are no biomarkers to help predict in which patients acute low back pain (LBP) will transform into chronic low back pain (CLBP). Human variability and different common comorbidities complicate the picture and make stratification of patients into correct subgroups difficult. However, drugs act by targeting specific molecular pathways and are therefore efficient only in a subgroup of patients sharing common molecular pathology and common genetics. Both CLBP and disc degeneration are known to be heritable. Little investigation has taken place for genetic variants in CLBP. The main aim of this trial is to identify "omics biomarkers" associated with the transition from acute (single episode of low back pain) to persistent/chronic LBP (pain lasting more than 12 weeks).

DETAILED DESCRIPTION:
Investigators will link and relate clinical data to a multiple "omics" analysis in patients developing persistent chronic symptoms (defined as pain that persists 3 months or more), after an episode of acute LBP. The development of persistent chronic pain will be assessed at 3 months after the acute episode.

"OMIC" biomarkers investigated will be genetics, epigenetics, glycomics and activomic.

Genetics through genome wide association studies (GWAS) has already obtained important results in pain research; however concerning low back pain, there is not yet suitable genotype-phenotype correlations helpful to stratify patients.

Epigenetic regulation is a universal tool that higher organisms use to adapt to changes in the environment. While environmental factors, such as diet influence enzymatic processes only while they are directly present, their prolonged effects can be achieved through the cell memory of epigenetic marks. Various elements of the membrane signal transduction system were reported to be regulated by epigenetic mechanisms.

Glycomics is an emerging field that has recently been identified as a priority for the next decade by the US National Academies of Science. Many common complex diseases will be associated with specific changes in glycan structures. In addition, common genetic polymorphisms influencing glycosylation and consequent differences in glycome composition could be important diagnostic and prognostic markers. The first studies reporting protein glycosylation in large human population samples have been recently published by partners in the consortium. Reliable identification of valid associations between specific glyco-phenotypes and predisposition for the development or progression of a specific disease requires analysis of thousands of patients.

Activomics: combines data about enzymatic activity of numerous numerous post-translational modification proteins in an integrated model which provides dynamic characterization of the current state of an organism. In this project information about numerous proteases, kinases, phosphatases and glycosidases will be collected and used to complement the existing phenotype information.

"Omics" data will be compared stratifying population according to pain characteristics, pain intensity, response to treatment and duration of pain. In a subgroup of patients, "omics" data will be compared stratifying population according to pain pathophysiology: discogenic pain, spinal stenosis, facet joint pain, sacroiliac joint pain, low back pain with radicular pain (radicular pain not predominant) and widespread low back pain.

ELIGIBILITY:
Inclusion Criteria:

* age: older than 18;
* acute episode of pain between the costal margins and gluteal fold, with or without symptoms into one or both legs lasting less than 6 weeks;
* written informed consent signed;
* Caucasian ancestry

Exclusion Criteria:

* evidence of clinically unstable disease;
* severe psychiatric disorder (excluding mild depression) or mental impairment;
* history (in the last 6 months) of persistent chronic low back pain or acute LBP episodes
* recent history (< 1 year) of spinal fracture;
* pain in the back due to spinal tumor or infection;
* pregnancy;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each clinical centre will identify patients with an episode of acute LBP, with or without irradiation, referred from primary care physicians, orthopaedic specialists or directly selected in the emergency room (accessing hospital for acute low back pain).
  The enrolment will be competitive among the participating clinical centres.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Genetic outcome | 54 months
  To investigate the associations between genetic factors and the development of persistent chronic LBP, in patients developing persistent chronic symptoms (defined as pain that persists 3 months or more), after an episode of acute LBP. The development of persistent chronic pain will be assessed at 3 months after the acute episode.
  Existing and newly generated GWAs will be analyzed and their possible correlation with the risk of pain becoming persistent chronic will be detected in a wide, international population of caucasian ancestry.

SECONDARY OUTCOMES:
Glycomic and Activomic outcome | 54 months
  Recognize Glycomic and Activomic data associated with patients who develop CLBP compared to patients who do not develop CLBP after an episode of acute LBP. The sample size will better defined after the first interim analysis of first 400 patients.
Epigenetic outcome | 54 months
  Investigators will identify CpG methylation patterns that may be associated with the development and maintenance of persistent chronic LBP pain after an episode of acute LBP in the first 200 patients who develop CLBP and first 200 patients who will not develop it.
  In the same cohort of 400 patients, investigators will analyze microRNAs (miRNAs) to investigate their role in predicting risk of persistent chronic pain after acute episode, opioid tolerance and response to therapy after the beginning of opioid therapy.
Next-generation sequencing outcome | 54 months
  Investigators will detect rare variants with strong or modest effects on LBP symptoms and response to therapy using next generation sequencing of candidate genes in 200 incident cases with persistent chronic pain and 200 controls. In particular, investigators will analyze new genetic variants that may impact on intervertebral disc stability, new variants modifying inflammation, variants of pain signalling, new variants in genes encoding analgesic drug metabolism and other genes from literature search.
Stratification based on pain characteristics | 54 months
  "Omics" data will be compared stratifying our population according to pain characteristics, pain intensity, response to treatment and duration of pain.
Stratification based on pain pathophysiology | 54 months
  In a subgroup of patients, "omics" data will be compared stratifying our population according to pain pathophysiology: discogenic pain, spinal stenosis, facet joint pain, sacroiliac joint pain, low back pain with radicular pain (radicular pain not predominant) and widespread low back pain.
Stratification based on 6 months follow-up | 54 months
  "Omics" data will be also compared stratifying our population according to the persistence of pain at 6 months despite receiving a treatment following current guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: MASSIMO ALLEGRI, MD, Principal Investigator — Pain Therapy Service Azienda Ospedaliera Universitaria Parma Italy
Locations (7):
- The Center for Clinical Research (CPI), Winston-Salem, North Carolina, United States
- Edith Cowan University (ECU), Perth, Australia
- Multidisciplinary Pain Centre, Hospital Oost-Limburg (ZOL), Genk, Belgium
- "St.Catharine" Orthopedics, Surgery, Neurology and Physical Medicine and Rehabilitation Specialty Hospital (St-Cat), Zabok, Croatia
- Italy (2):
  - Anesthesia and Pain Therapy Department, Università degli Studi di Parma (UNIPR), Parma
  - Fondazione IRCCS Policlinico San Matteo (OSM), Pavia
- King's College London (KCL), London, United Kingdom